CLINICAL TRIAL: NCT01644175
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of SAR236553/REGN727 in High Cardiovascular Risk Patients With Hypercholesterolemia Not Adequately Controlled With Their Lipid-Modifying Therapy
Brief Title: Efficacy and Safety of Alirocumab (SAR236553/REGN727) Versus Placebo on Top of Lipid-Modifying Therapy in Patients With High Cardiovascular Risk and Hypercholesterolemia (ODYSSEY COMBO I)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC11568; U1111-1121-4356 (Other: UTN)
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Q2W (Placebo Comparator): Placebo (for alirocumab) every 2 weeks (Q2W) added to stable Lipid-Modifying Therapy (LMT) for 52 weeks.
  Interventions: Drug: Placebo (for alirocumab); Drug: Lipid-Modifying Therapy (LMT)
- Alirocumab (Experimental): Alirocumab 75 mg Q2W added to stable LMT for 52 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) at Week 8.
  Interventions: Drug: Alirocumab; Drug: Lipid-Modifying Therapy (LMT)

INTERVENTIONS:
Drug: Placebo (for alirocumab) — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with a disposable auto-injector (also known as pre-filled pen).
  Arms: Placebo Q2W
Drug: Alirocumab — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with a disposable auto-injector (also known as pre-filled pen).
  Other Names: SAR236553; REGN727
  Arms: Alirocumab
Drug: Lipid-Modifying Therapy (LMT) — Statin (rosuvastatin, simvastatin or atorvastatin) at stable dose with or without other LMT as clinically indicated.

SUMMARY:
Alirocumab (SAR236553/REGN727) is a fully human monoclonal antibody that binds proprotein convertase subtilisin/kexin type 9 (PCSK9).

Primary Objective of the study:

* To demonstrate the reduction of low-density lipoprotein cholesterol (LDL-C) by alirocumab as add-on therapy to stable maximally tolerated daily statin therapy with or without other lipid-modifying therapy (LMT) in comparison with placebo after 24 weeks of treatment in high cardiovascular (CV) risk participants with hypercholesterolemia

Secondary Objectives:

* To evaluate the effect of alirocumab in comparison with placebo on LDL-C at other time points
* To evaluate the effect of alirocumab on other lipid parameters
* To evaluate the safety and tolerability of alirocumab

DETAILED DESCRIPTION:
The maximum study duration was 62 weeks per participant, including a 2-week screening period, 52-week randomized treatment period, and 8-week follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Participants with hypercholesterolemia and established coronary heart disease (CHD) or CHD risk equivalents who were not adequately controlled with a maximally tolerated daily dose of statin with or without other LMT, both at stable dose for at least 4 weeks to 6 weeks prior to screening (Week -2)

Exclusion criteria:

* Age <18 or legal age of adulthood, whichever was greater
* Participants without established CHD or CHD risk equivalent
* LDL-C <70 mg/dL (<1.81 mmol/L) and participants with a history of documented cardiovascular disease
* LDL-C <100 mg/dL (<2.59 mmol/L) and participants without a history of documented cardiovascular disease
* Not on a stable dose of LMT (including statin) for at least 4 weeks and/or fenofibrate for at least 6 weeks, as applicable, prior to the screening visit (Week -2) and from screening to randomization
* Fasting serum triglycerides > 400 mg/dL (>4.52 mmol/L)

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (76):
- United States (76):
  - Investigational Site Number 840857, Birmingham, Alabama
  - Investigational Site Number 840891, Mobile, Alabama
  - Investigational Site Number 840876, Montgomery, Alabama
  - Investigational Site Number 840865, Glendale, Arizona
  - Investigational Site Number 840826, Jonesboro, Arkansas
  - Investigational Site Number 840870, Burbank, California
  - Investigational Site Number 840851, Los Angeles, California
  - Investigational Site Number 840845, Los Gatos, California
  - Investigational Site Number 840844, Sacramento, California
  - Investigational Site Number 840801, San Jose, California
  - Investigational Site Number 840886, Tarzana, California
  - Investigational Site Number 840862, Torrance, California
  - Investigational Site Number 840893, Vista, California
  - Investigational Site Number 840867, Boca Raton, Florida
  - Investigational Site Number 840884, Boynton Beach, Florida
  - Investigational Site Number 840836, Clearwater, Florida
  - Investigational Site Number 840866, Coral Gables, Florida
  - Investigational Site Number 840895, Fort Lauderdale, Florida
  - Investigational Site Number 840820, Hialeah, Florida
  - Investigational Site Number 840805, Miami, Florida
  - Investigational Site Number 840811, Oviedo, Florida
  - Investigational Site Number 840881, Port Orange, Florida
  - Investigational Site Number 840816, West Palm Beach, Florida
  - Investigational Site Number 840850, Columbus, Georgia
  - Investigational Site Number 840840, Eagle, Idaho
  - Investigational Site Number 840842, Chicago, Illinois
  - Investigational Site Number 840898, Evanston, Illinois
  - Investigational Site Number 840847, Morton, Illinois
  - Investigational Site Number 840896, Indianapolis, Indiana
  - Investigational Site Number 840894, Michigan City, Indiana
  - Investigational Site Number 840838, Mishawaka, Indiana
  - Investigational Site Number 840823, Paducah, Kentucky
  - Investigational Site Number 840858, Eunice, Louisiana
  - Investigational Site Number 840802, New Orleans, Louisiana
  - Investigational Site Number 840855, Salisbury, Massachusetts
  - Investigational Site Number 840890, Battle Creek, Michigan
  - Investigational Site Number 840832, Southfield, Michigan
  - Investigational Site Number 840839, Edina, Minnesota
  - Investigational Site Number 840888, Minneapolis, Minnesota
  - Investigational Site Number 840837, Port Gibson, Mississippi
  - Investigational Site Number 840814, Jefferson City, Missouri
  - Investigational Site Number 840833, Sparks, Nevada
  - Investigational Site Number 840817, Newington, New Hampshire
  - Investigational Site Number 840853, New Windsor, New York
  - Investigational Site Number 840822, Rochester, New York
  - Investigational Site Number 840824, Cary, North Carolina
  - Investigational Site Number 840880, Smithfield, North Carolina
  - Investigational Site Number 840502, Winston-Salem, North Carolina
  - Investigational Site Number 840852, Winston-Salem, North Carolina
  - Investigational Site Number 840846, Cincinnati, Ohio
  - Investigational Site Number 840899, Cincinnati, Ohio
  - Investigational Site Number 840831, Columbus, Ohio
  - Investigational Site Number 840860, Kettering, Ohio
  - Investigational Site Number 840809, Willoughby Hills, Ohio
  - Investigational Site Number 840818, Norman, Oklahoma
  - Investigational Site Number 840812, Eugene, Oregon
  - Investigational Site Number 840803, Downington, Pennsylvania
  - Investigational Site Number 840869, Philadelphia, Pennsylvania
  - Investigational Site Number 840825, Pittsburgh, Pennsylvania
  - Investigational Site Number 840872, Anderson, South Carolina
  - Investigational Site Number 840885, Charleston, South Carolina
  - Investigational Site Number 840813, Greer, South Carolina
  - Investigational Site Number 840827, Mt. Pleasant, South Carolina
  - Investigational Site Number 840868, Corpus Christi, Texas
  - Investigational Site Number 840877, Houston, Texas
  - Investigational Site Number 840841, Houston, Texas
  - Investigational Site Number 840830, San Antonio, Texas
  - Investigational Site Number 840854, San Antonio, Texas
  - Investigational Site Number 840883, San Antonio, Texas
  - Investigational Site Number 840889, Tomball, Texas
  - Investigational Site Number 840878, Bountiful, Utah
  - Investigational Site Number 840819, Orem, Utah
  - Investigational Site Number 840863, Salt Lake City, Utah
  - Investigational Site Number 840804, Manassas, Virginia
  - Investigational Site Number 840882, Norfolk, Virginia
  - Investigational Site Number 840810, Weber City, Virginia

REFERENCES:
- [Background] Colhoun HM, Robinson JG, Farnier M, Cariou B, Blom D, Kereiakes DJ, Lorenzato C, Pordy R, Chaudhari U. Efficacy and safety of alirocumab, a fully human PCSK9 monoclonal antibody, in high cardiovascular risk patients with poorly controlled hypercholesterolemia on maximally tolerated doses of statins: rationale and design of the ODYSSEY COMBO I and II trials. BMC Cardiovasc Disord. 2014 Sep 20;14:121. doi: 10.1186/1471-2261-14-121. PMID 25240705
- [Result] Kereiakes DJ, Robinson JG, Cannon CP, Lorenzato C, Pordy R, Chaudhari U, Colhoun HM. Efficacy and safety of the proprotein convertase subtilisin/kexin type 9 inhibitor alirocumab among high cardiovascular risk patients on maximally tolerated statin therapy: The ODYSSEY COMBO I study. Am Heart J. 2015 Jun;169(6):906-915.e13. doi: 10.1016/j.ahj.2015.03.004. Epub 2015 Mar 13. PMID 26027630
- [Derived] Mahmood T, Minnier J, Ito MK, Li QH, Koren A, Kam IW, Fazio S, Shapiro MD. Discordant responses of plasma low-density lipoprotein cholesterol and lipoprotein(a) to alirocumab: A pooled analysis from 10 ODYSSEY Phase 3 studies. Eur J Prev Cardiol. 2021 Jul 23;28(8):816-822. doi: 10.1177/2047487320915803. Epub 2020 Apr 10. PMID 34298554
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Ray KK, Ginsberg HN, Davidson MH, Pordy R, Bessac L, Minini P, Eckel RH, Cannon CP. Reductions in Atherogenic Lipids and Major Cardiovascular Events: A Pooled Analysis of 10 ODYSSEY Trials Comparing Alirocumab With Control. Circulation. 2016 Dec 13;134(24):1931-1943. doi: 10.1161/CIRCULATIONAHA.116.024604. Epub 2016 Oct 24. PMID 27777279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 76 centers in the United States of America. Overall, 640 participants were screened between July 2012 and February 2013, 324 of whom were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified according to prior history of myocardial infarction (MI) or ischemic stroke, and intensity of statin treatment. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 1:2 ratio (placebo: alirocumab) after confirmation of selection criteria. 316 participants were randomized.
Groups:
- Placebo Q2W: Placebo (for alirocumab) subcutaneous (SC) injection every 2 weeks (Q2W) added to stable Lipid-Modifying Therapy (LMT) for 52 weeks.
- Alirocumab 75/150 mg Q2W: Alirocumab 75 mg SC injection Q2W added to stable LMT for 52 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) at Week 8.
Period: Overall Study
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Started | 107 (Randomized) | 209 (Randomized)
Treated | 107 | 207
Completed | 75 | 156
Not Completed | 32 | 53
Not completed — Randomized But Not Treated | 0 | 2
Not completed — Adverse Event | 8 | 13
Not completed — Death | 1 | 2
Not completed — Poor compliance to protocol | 9 | 10
Not completed — Physician Decision | 1 | 2
Not completed — Participant Moved | 1 | 2
Not completed — Consent withdrawn by participant | 3 | 4
Not completed — Related to Autoinjector Administration | 2 | 1
Not completed — Last visit outside protocol visit window | 4 | 11
Not completed — Selection criteria finally not met | 0 | 1
Not completed — Site closure | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other than specified above | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo Q2W: Placebo (for alirocumab) SC injection Q2W added to stable LMT for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W | Total
Number analyzed (Participants) | 107 | 209 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (8.8) | 63.0 (9.5) | 63.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 78 | 108
  Male | 77 | 131 | 208
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] — Calculated LDL-C in mmol/L from Friedewald formula (LDL cholesterol = Total cholesterol - HDL cholesterol - [Triglyceride/2.2]).
  mmol/L | 2.746 (0.915) | 2.595 (0.764) | 2.646 (0.820)
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C in mg/dL from Friedewald formula (LDL cholesterol = Total cholesterol - HDL cholesterol - [Triglyceride/5]).
  mg/dL | 106.0 (35.3) | 100.2 (29.5) | 102.2 (31.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent-to-Treat (ITT) Analysis
Description: Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 52
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | -2.3 (2.7) | -48.2 (1.9)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; Alirocumab group was compared to placebo group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -45.9, 95% CI 2-sided [-52.5 to -39.3] — Alirocumab vs. placebo

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection) (on-treatment analysis).
Time Frame: From Baseline to Week 52
Population: Modified ITT (mITT) population: all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 105 | 204
percent change | -0.8 (2.6) | -50.7 (1.9)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance was ≤ 0.05; LS Mean Difference = -49.9, 95% CI 2-sided [-56.2 to -43.6] — Alirocumab vs. placebo

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | 1.1 (2.5) | -46.3 (1.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -47.4, 95% CI 2-sided [-53.6 to -41.3] — Alirocumab vs. placebo

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 105 | 204
percent change | 1.7 (2.5) | -47.6 (1.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -49.3, 95% CI 2-sided [-55.3 to -43.3] — Alirocumab vs. placebo

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment (Apo B ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 96 | 185
percent change | -0.9 (2.3) | -36.7 (1.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -35.8, 95% CI 2-sided [-41.3 to -30.3] — Alirocumab vs. placebo

6. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 - On-treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: Participants of the mITT population with one baseline and at least one post-baseline Apo B value on-treatment (Apo B mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 93 | 181
percent change | -0.4 (2.3) | -37.9 (1.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤0.05; LS Mean Difference = -37.5, 95% CI 2-sided [-43.0 to -32.0] — Alirocumab vs. placebo

7. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | -1.6 (2.5) | -39.1 (1.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -37.5, 95% CI 2-sided [-43.5 to -31.4] — Alirocumab vs. placebo

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - On-treatment Analysis
Description: as for outcome 6
Time Frame: From Baseline to Week 52
Population: Participants of the mITT population with one baseline and at least one post-baseline non-HDL-C value on-treatment (non-HDL-C mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 105 | 204
percent change | -0.5 (2.5) | -40.9 (1.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -40.4, 95% CI 2-sided [-46.4 to -34.4] — Alirocumab vs. placebo

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Total-C value on- or off-treatment (Total-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | -2.9 (1.8) | -27.9 (1.3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -25.0, 95% CI 2-sided [-29.3 to -20.7] — Alirocumab vs. placebo

10. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 52
Population: Apo B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 96 | 185
percent change | 3.4 (2.3) | -34.8 (1.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -38.2, 95% CI 2-sided [-43.7 to -32.7] — Alirocumab vs. placebo

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 52
Population: Non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | 2.6 (2.6) | -37.4 (1.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -40.1, 95% CI 2-sided [-46.2 to -33.9] — Alirocumab vs. placebo

12. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 52
Population: Total-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | 0.9 (2.0) | -25.4 (1.4)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -26.4, 95% CI 2-sided [-31.1 to -21.7] — Alirocumab vs. placebo

13. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 52 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | 0.5 (3.6) | -42.5 (2.5)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -43.0, 95% CI 2-sided [-51.6 to -34.3] — Alirocumab vs. placebo

14. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 were obtained from multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: Up to Week 52
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percentage of participants | 9.0 | 75.0
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 38.5, 95% CI 2-sided [16.5 to 89.8] — Alirocumab vs. placebo

15. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-treatment Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach model including available post-baseline on-treatment data from Week 4 to Week 52 i.e. up to 21 days after last injection.
Time Frame: Up to Week 52
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 105 | 204
percentage of participants | 8.0 | 77.5
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 50.0, 95% CI 2-sided [20.6 to 121.0] — Alirocumab vs. placebo

16. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 were obtained from multiple imputation approach followed by robust regression model for handling of missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: From baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | -5.9 (2.8) | -20.5 (2.0)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -14.6, 95% CI 2-sided [-21.3 to -7.9] — Alirocumab vs. placebo

17. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | -3.8 (1.5) | 3.5 (1.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 7.3, 95% CI 2-sided [3.6 to 11.0] — Alirocumab vs. placebo

18. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from multiple imputation approach followed be robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | -5.4 (3.2) | -6.0 (2.3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75/150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8699, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -0.6, 95% CI 2-sided [-8.3 to 7.0] — Alirocumab vs. placebo

19. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo A-1 value on- or off-treatment (Apo A-1 ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 96 | 185
percent change | -2.5 (1.2) | 3.3 (0.9)

20. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12- ITT Analysis
Description: Adjusted means and standard errors at Week 12 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | 0.0 (2.7) | -19.7 (1.9)

21. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 52
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | -2.4 (1.4) | 6.7 (1.0)

22. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from multiple imputation approach followed by a robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 106 | 205
percent change | 3.0 (2.9) | -11.3 (2.0)

23. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 52
Population: Apo A-1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75/150 mg Q2W
Number analyzed (Participants) | 96 | 185
percent change | -1.8 (1.3) | 3.8 (0.9)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 60 post-treatment follow-up visit) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'treatment emergent period' (the time from the first dose of study drug up to the last dose of study drug +70 days).
Groups:
- Placebo Q2W: Participants exposed to placebo (for alirocumab) SC injection Q2W added to stable LMT (mean exposition of 45 weeks).
- Alirocumab 75 /up to 150 mg Q2W: Participants exposed to alirocumab 75 mg /up to 150 mg SC injection Q2W added to stable LMT (mean exposition of 46 weeks).
Arm/Group | Placebo Q2W | Alirocumab 75 /up to 150 mg Q2W
Serious Adverse Events (participants affected / at risk) | 14/107 | 26/207
Other Adverse Events (participants affected / at risk) | 31/107 | 72/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=107) | Alirocumab 75 /up to 150 mg Q2W (N=207)
Bronchitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 0
Sudden cardiac death (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Tooth injury (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=107) | Alirocumab 75 /up to 150 mg Q2W (N=207)
Upper respiratory tract infection (Infections and infestations) | 11 | 16
Nasopharyngitis (Infections and infestations) | 5 | 15
Urinary tract infection (Infections and infestations) | 4 | 13
Sinusitis (Infections and infestations) | 4 | 11
Dizziness (Nervous system disorders) | 6 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 8
Injection site reaction (General disorders) | 3 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.